CLINICAL TRIAL: NCT05757024
Title: Effect Of High Power Laser Therapy On Radiotherapy Induced Trismus In Head And Neck Cancer Patients
Brief Title: Effect Of High Power Laser On Radiotherapy Induced Trismus.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Hassan Abdel Twab Hussein, doctor of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012004161
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Trismus
MeSH Terms: conditions — Trismus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): study group receive high power laser therapy in combination with conventional tempromandibular joint exercises.
  Interventions: Device: high power laser therapy
- control group (Active Comparator): control group receive traditional tempromadibular joint exercises.
  Interventions: Device: high power laser therapy

INTERVENTIONS:
Device: high power laser therapy — m6 laser therapy of ASA company with multilocked wave system and synchronized emission wave lengths 808 and 905 wave lengths
  Other Names: conventional tempromandibular joint exercises

SUMMARY:
this study Randomized controlled study will be conducted to study (the effect of high power laser therapy on radiotherapy induced trismus in head and neck cancer patients).

the study group will receive high power laser therapy in combination with conventional tempromandibular joint exercises.

the control group will receive conventional tempromandibular joint exercises.

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer patients who complain of decreased mouth opening and received or receiving radiotherapy.
* patients who complain from pain and inflammation in the tempromandibular joint due to radiotherapy.
* radiotherapy should be above 40 GY.
* patient ages between 20 to 65 years old.

Exclusion Criteria:

* patients with poor general health.
* patients with difficulties in filling questionnaire.
* patients who are complaining of other tempomandibular problems other than trismus such as (disc discplacement and trumatic mandibular fractures.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
pain level | one month (4 weeks)
  visual analogue scale
mouth opening | one month (4 weeks)
  verneir caliper

SECONDARY OUTCOMES:
quality of life improvement | one month (4 weeks)
  Washington quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Hussein Elgendy, proffessor, Study Director — Faculty of physiacl therapy cairo university
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
study limitations and recommendations

REFERENCES:
- [Result] Zecha JA, Raber-Durlacher JE, Nair RG, Epstein JB, Elad S, Hamblin MR, Barasch A, Migliorati CA, Milstein DM, Genot MT, Lansaat L, van der Brink R, Arnabat-Dominguez J, van der Molen L, Jacobi I, van Diessen J, de Lange J, Smeele LE, Schubert MM, Bensadoun RJ. Low-level laser therapy/photobiomodulation in the management of side effects of chemoradiation therapy in head and neck cancer: part 2: proposed applications and treatment protocols. Support Care Cancer. 2016 Jun;24(6):2793-805. doi: 10.1007/s00520-016-3153-y. Epub 2016 Mar 17. PMID 26984249
- [Result] Borges, Marcela Maria Fontes, et al.